CLINICAL TRIAL: NCT02000297
Title: Outcome Comparison of Allogenic Cancellous Bone and a New Synthetic Bone Substitute (geneX®) in Filling the Bone Defect Created With Medial Open Wedge High Tibial Osteotomy
Brief Title: Outcome Comparison of Allograft and Synthetic Bone Substitute in High Tibial Osteotomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Tae Kyun Kim, Direcor, Joint reconstruction center, SNUBH, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B-1309/220-005
Record Dates: First submitted 2013-11-11; First posted 2013-12-04 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; High tibial osteotomy; Calcium phosphate; Calcium sulfate
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Allogenic bone graft group (Active Comparator): Patients in this arm is treated with allogenic bone graft to fill the bone defect created with medial open wedge high tibial osteotomy
  Interventions: Procedure: Allogenic bone graft
- Synthetic bone substitute (geneX®) group (Experimental): Patients in this arm is treated with synthetic bone substitute(geneX®) to fill the bone defect created with medial open wedge high tibial osteotomy
  Interventions: Procedure: Synthetic bone substitute (geneX®)

INTERVENTIONS:
Procedure: Allogenic bone graft — Patients in this arm is treated with allogenic bone graft to fill the bone defect created with medial open wedge high tibial osteotomy
  Arms: Allogenic bone graft group
Procedure: Synthetic bone substitute (geneX®) — Patients in this arm is treated with synthetic bone substitute (geneX®) to fill the bone defect created with medial open wedge high tibial osteotomy
  Arms: Synthetic bone substitute (geneX®) group

SUMMARY:
This study is conducted to determine whether a new synthetic bone substitute is better than allogenic bone graft for addressing bone defect in medial open wedge high tibial osteotomy in terms of postoperative pain, postoperative bleeding, operation time and bone healing. The investigators hypothesized the new synthetic bone substitute would bring better outcomes in the outcome variables mentioned above.

DETAILED DESCRIPTION:
High tibial osteotomy is a well-established treatment option for the young patients (aged 40~55years) with knee osteoarthritis which is confined in medial compartment of the knee. Classical technique was lateral closing wedge osteotomy, but recently medial open wedge osteotomy has gained popularity with the advent of new fixation devices and refined surgical techniques. The surgeon can correct the deformity more precisely in both coronal and sagittal planes simultaneously with medial opening technique. And it can avoid complications associated with lateral closing technique like tibial shaft offset or peroneal nerve palsy. But medial opening technique inevitably creates large bone defect, which has to be addressed to avoid complications like loss of correction or delayed/non-union. Autologous bone is widely accepted as a standard for filling bone defects, but its supply is limited and harvesting autologous bone adds to surgical morbidity like bleeding, pain or fracture at the donor site. Therefore, there has been much effort to find materials to substitute autologous bone. Many studies reported the results of using allogenic bone for addressing bone defects and most of them showed favorable results. But some allogenic bone products are cumbersome to process to make it fit to the defect, and there are potential risk of disease transmission, if the products are not properly treated. Bone cements of several different composition has been developed and when used for filling bone defect, they also showed good results in general. Recently, a new synthetic bone substitute based on calcium phosphate and calcium sulfate (geneX®, Biocomposites Co.,Ltd.) has been introduced and is commercially available. While providing initial mechanical strength, its calcium sulfate component is rapidly absorbed to provide space for new bone ingrowth and its surface is made to negatively charged, which helps accelerate new bone formation. It is provided as an injectable paste, which is easier to handle than allogenic bone, so it may help reduce operation time. With these theoretical advantages, there are some anecdotal reports that patients treated with geneX® presented less postoperative pain and bleeding than patients treated with allogenic bone graft. Therefore, we conducted this study to determine whether the new synthetic bone substitute (geneX®) is better than allogenic bone for addressing bone defect created in medial open wedge high tibial osteotomy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary osteoarthritis of the knee which is confined to medial compartment
* Scheduled for high tibial osteotomy
* Written signed consent available

Exclusion Criteria:

* Patients who refuse to participate in the study
* Previous history of major orthopedic surgery around the operating knee
* Congenital anomaly involving proximal tibia
* Revision high tibial osteotomy
* Patients who is receiving another major knee surgery simultaneously with high tibial osteotomy at the same knee

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-10; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Temporal change of postoperative pain | from 2 days after surgery to 12 months after surgery
  Pain on operation site is measured on a 0-to-10 visual analogue scale(VAS) and 5-point Likert scale (0.no pain, 1.slight pain, 2.moderate pain, 3.severe pain, 4.extreme pain).
  Initial postoperative pain will be recorded on postoperative day 2. After discharge from hospital (on postoperative day 2, on average), patients will visit outpatient department on 2weeks, 6weeks, 3months, 6months, 12months after surgery and pain measurements on each visit will be recorded.

SECONDARY OUTCOMES:
Pre&postoperative Hemoglobin level | on admission (preop.), postoperative day 2 (postop.)
  Preoperative hemoglobin level is measured when the patient is admitted to the hospital for surgery and postoperative level is measured on postoperative day 2. The differences between values will be calculated.
Total operation time | from skin incision to deflation of tourniquet
  Total operation time is defined as the time interval between skin incision and deflation of tourniquet (thigh tourniquet used in the operation to provide bloodless surgical field). Measured in minutes.
Temporal change of weight bearing status | from 2 weeks after surgery to 12 months after surgery
  As a proxy variable of bone healing status, whether the patient can bear weight on operated knee is measured on a 3 point scale (1.full weight bearing, 2.partial weight bearing, 3.no weight bearing)
  Patients will visit outpatient department on 2weeks, 6weeks, 3months, 6months, 12months after surgery and weight bearing status on each visit will be recorded.
Temporal change of pain with weight bearing | from 2 weeks after surgery to 12 months after surgery
  As a proxy variable of bone healing status, pain with weight bearing is measured on a 0-to-10 visual analogue scale(VAS) and 5-point Likert scale (0.no pain, 1.slight pain, 2.moderate pain, 3.severe pain, 4.extreme pain)
  Patients will visit outpatient department on 2weeks, 6weeks, 3months, 6months, 12months after surgery and pain with weight bearing on each visit will be recorded.
Amount of drainage | from the end of surgery until drain removal, which is anticipated on postoperative day 1 or 2
  Total amount of drainage (in milliliters) from indwelling drain located in operative site, until its removal.
Working time for bone defect filling | from the start of processing allograft or synthetic bone substitute to finish filling bone defect
  Time required to fill the bone defect (from the start of processing either allogenic bone graft or synthetic bone substitute to completely finish filling the defect. Measured in seconds.
Temporal progression of bone healing on X-rays | from 3 months after surgery to 12months after surgery
  Two independent investigators assess the progression of bone healing status on X-rays and the agreement between investigators will be measured. Bone healing status is assessed based on 3 point scale. (1. union not achieved yet, 2. partial union achieved, 3. complete union achieved)
  Patients will visit outpatient department on 2weeks, 6weeks, 3months, 6months, 12months after surgery and bone healing status on X-rays will be recorded on 3months, 6months and 12months after surgery.

OTHER OUTCOMES:
Amount of transfusion | from the start of operation until discharge of the patient from hospital (which is anticipated on postoperative day 2 on average)
  Amount of transfusion during patient's hospital stay, if any, is measured in packs.
Postoperative complications | from the date of operation to the date of occurence of any complications, assessed up to 12 months after surgery
  When an event of postoperative complication occurs, it is recorded with postoperative date.

CONTACTS AND LOCATIONS:
Overall Officials: Tae Kyun Kim, MD, PhD, Principal Investigator — Joint Reconstruction Center, Seoul National University Bundang Hospital
Locations (1):
- Joint Reconstruction Center, Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea